CLINICAL TRIAL: NCT00020475
Title: Phase II Study of gp100:209-217 (210M) Antigen and MART-1:26-35 (27L) Antigen Emulsified in Montanide ISA-51 in Patients With Metastatic Ocular Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma of the Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068514; NCI-01-C-0074; NCI-2910; NCT00009516 (obsolete NCT alias)
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Extraocular Extension Melanoma; Recurrent Intraocular Melanoma
Keywords: adult solid tumor; body system/site cancer; cancer; extraocular extension melanoma; eye cancer; intraocular melanoma; recurrent intraocular melanoma; solid tumor; stage, intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Neoplasms; Eye Neoplasms | interventions — Interleukin-2; MART-1 Antigen; montanide ISA 51

INTERVENTIONS:
Drug: gp100 antigen
Drug: interleukin-2
Drug: MART-1 antigen
Drug: Montanide ISA-51

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Combining vaccine therapy with interleukin-2 may be a more effective treatment for metastatic melanoma of the eye.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy and interleukin-2 in treating patients who have metastatic melanoma of the eye.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical response in patients with metastatic ocular melanoma treated with gp100:209-217 (210M) antigen and MART-1:26-35 (27L) antigen emulsified in Montanide ISA-51.

II. Determine the clinical benefit of interleukin-2 in combination with this vaccine in these patients.

PROTOCOL OUTLINE: Patients receive vaccine subcutaneously once weekly. Treatment repeats every 4 weeks for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with progressive disease may receive vaccine SC on day 1 followed by interleukin-2 IV over 15 minutes every 8 hours for a maximum of 12 doses. Treatment repeats every 3 weeks for at least 4 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL:

A total of 15-25 patients will be accrued for this study within 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnosis of metastatic ocular melanoma Progressive disease Measurable disease HLA-A*201 positive --Prior/Concurrent Therapy-- Biologic therapy: At least 3 weeks since prior biologic therapy Chemotherapy: At least 3 weeks since prior chemotherapy Endocrine therapy: At least 3 weeks since prior endocrine therapy No concurrent steroid therapy Radiotherapy: At least 3 weeks since prior radiotherapy Surgery: Not specified --Patient Characteristics-- Age: 16 and over Performance status: ECOG 0-2 Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 90,000/mm3 No coagulation disorders Hepatic: Bilirubin no greater than 2.0 mg/dL AST/ALT less than 3 times normal Hepatitis B surface antigen negative Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No major cardiovascular illness For interleukin-2 (IL-2) therapy: No cardiac ischemia No myocardial infarction No cardiac arrhythmias Pulmonary: No major respiratory system illness For IL-2 therapy: No obstructive or restrictive pulmonary disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active systemic infection No autoimmune disease No primary or secondary immunodeficiency by abnormal lymphocyte counts or presence of opportunistic infection

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-02; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco M. Marincola, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States